CLINICAL TRIAL: NCT04172896
Title: Comparison of Vaginal Intraperitoneal and Extraperitoneal Uterosacral Ligament Suspensions for Post-Hysterectomy Vaginal Vault Prolapse: A Randomized Clinical Trial
Brief Title: Intraperitoneal and Extraperitoneal Uterosacral Ligament Suspensions for Post-Hysterectomy Vaginal Vault Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Danny Mounir, Clinical Fellow, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00022633
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Vaginal Vault Prolapse; Post-Hysterectomy Vaginal Vault Prolapse; Prolapse, Vaginal
Keywords: Pelvic Reconstructive Surgery; Prolapse Surgery
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel design. Participants will be randomly assigned to either vaginal intraperitoneal or extraperitoneal uterosacral ligament suspension.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraperitoneal Group (Active Comparator): Vaginal intraperitoneal uterosacral ligament suspension group
  Interventions: Procedure: Intraperitoneal Uterosacral Ligament Suspension
- Extraperitoneal Group (Active Comparator): Vaginal extraperitoneal uterosacral ligament suspension group
  Interventions: Procedure: Extraperitoneal Uterosacral Ligament Suspension

INTERVENTIONS:
Procedure: Intraperitoneal Uterosacral Ligament Suspension — Vaginal intraperitoneal uterosacral ligament suspension performed by transfixing the ligament, intraperitoneally, in the intermediate portion (at the level of or above ischial spine plane) with three delayed absorbable 0 sutures, performed bilaterally (three sutures per side; six sutures total).
  Arms: Intraperitoneal Group
Procedure: Extraperitoneal Uterosacral Ligament Suspension — Vaginal extraperitoneal uterosacral ligament suspension performed by transfixing the ligament, extraperitoneally, in the intermediate portion (at the level of or above ischial spine plane) using a suture capturing device with two delayed absorbable 0 sutures, performed bilaterally (two sutures per side; four sutures total).
  Arms: Extraperitoneal Group

SUMMARY:
Post-hysterectomy vaginal vault prolapse is a common pelvic floor disorder described as descent of the vaginal apex after hysterectomy. The incidence of post-hysterectomy vault prolapse has been reported to follow 11.6% of hysterectomies performed for prolapse and 1.8% for other benign diseases. The majority of surgical repairs to correct post-hysterectomy vault prolapse are approached via a transvaginal route. A common transvaginal procedure to correct vaginal vault prolapse is the uterosacral ligament suspension. Traditionally, the uterosacral ligaments have been accessed intraperitoneally to perform the vaginal suspension. More recently, an extraperitoneal approach has been utilized with good results. There is limited evidence comparing the the two approaches. Thus, the objectives of this study are to compare compare operative time, hospital stay, cost, surgical success, and other perioperative outcomes between the two approaches.

DETAILED DESCRIPTION:
This is a single-center, randomized, single-blind surgical trial of women with post-hysterectomy vaginal vault prolapse desiring surgical treatment. The purpose of this study is to compare outcomes of vaginal intraperitoneal uterosacral ligament suspensions and vaginal extraperitoneal uterosacral ligament suspensions for the treatment of post-hysterectomy vaginal vault prolapse. The primary objective will be to compare operative time between the two approaches. Secondary objectives of the trial will be to compare hospital stay, cost, surgical success, and other perioperative outcomes between the two approaches through 12 months using assessments at six weeks, six months, and twelve months.

The study will include subjects with stage 1-4 pelvic organ prolapse and descent of the vaginal apex at least ½ way into vaginal canal (defined as POPQ Point C ≥ -TVL/2) that desire vaginal surgical management for post-hysterectomy vaginal vault prolapse. Subjects enrolled into the trial will be randomized to either vaginal intraperitoneal or extraperitoneal uterosacral ligament suspension with a 1:1 allocation using a computer-generated randomization schedule. Patients will be blinded to their allocation. Patients in both groups will receive the same standard of care for vaginal procedures as it currently exists in out practice. This involves the standard anesthetics and opioid medications intraoperatively. Randomization will be revealed to the surgeons in the operating room once the patient is under general anesthesia.

Intraoperative data to be collected will include, operative time (minutes from surgical incision time to surgery end time), estimated blood loss (ml), intraoperative complications, and concurrent surgical procedures.

Preoperative and postoperative clinical measures to be collected will include POPQ examination points and scores from three validated questionnaires (Pelvic Floor Disability Index (PFDI-20) questionnaire, Pelvic Floor Impact Questionnaires (PFIQ-7) and the Pelvic and Incontinence Sexual Questionnaire (PISQ-12)). Postoperative clinical measures will be collected at six week, six month, and twelve month post-operative visits.

Surgical success or failure will be evaluated as a dichotomous composite outcome(objective measures (POPQ examination points) and subjective measures(validated questionnaires) at six week, six month, and twelve month post-operative visits.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 years of age or greater
* English speaking
* Stage 1 or greater post-hysterectomy vaginal vault prolapse
* Descent of vaginal apex at least ½ way into vaginal canal (defined as POPQ Point C ≥ -TVL/2)
* Vaginal surgery for prolapse is planned, including a vaginal apical suspension procedure

Exclusion Criteria:

* Non-English speaking or not able to provide informed consent
* Combined surgical cases with other surgical specialties
* Women unable to follow up postoperatively

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with post-hysterectomy vaginal vault prolapse
Enrollment: 34 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Operative time (minutes) | Day of surgery
  Minutes from surgical incision time to surgery end time

SECONDARY OUTCOMES:
Percent of participants with surgical "success" or "failure" as a dichotomous outcome at the 6 week postoperative visit | 6 week
  Surgical failure defined as any of the following: (1) apical descent greater than one-third of the total vaginal length or anterior or posterior vaginal wall beyond the hymen (2) retreatment for prolapse or (3) bothersome vaginal bulge symptoms as indicated by an positive response to either "Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?" or "Do you usually experience heaviness or dullness in the pelvic area?" in the Pelvic Floor Distress Inventory (PFDI-20), and any response other than "not at all" to the question "How much does this bother you?"
  A subject will be considered a surgical failure if any ONE of the criteria above is met. Otherwise, a subject will be considered a surgical success
Percent of participants with surgical "success" or "failure" as a dichotomous outcome at the 6 month postoperative visit | 6 month
  Surgical failure defined as any of the following: (1) apical descent greater than one-third of the total vaginal length or anterior or posterior vaginal wall beyond the hymen (2) retreatment for prolapse or (3) bothersome vaginal bulge symptoms as indicated by an positive response to either "Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?" or "Do you usually experience heaviness or dullness in the pelvic area?" in the Pelvic Floor Distress Inventory (PFDI-20), and any response other than "not at all" to the question "How much does this bother you?"
  A subject will be considered a surgical failure if any ONE of the criteria above is met. Otherwise, a subject will be considered a surgical success
Percent of participants with surgical "success" or "failure" as a dichotomous outcome at the 12 month postoperative visit | 12 month
  Surgical failure defined as any of the following: (1) apical descent greater than one-third of the total vaginal length or anterior or posterior vaginal wall beyond the hymen (2) retreatment for prolapse or (3) bothersome vaginal bulge symptoms as indicated by an positive response to either "Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?" or "Do you usually experience heaviness or dullness in the pelvic area?" in the Pelvic Floor Distress Inventory (PFDI-20), and any response other than "not at all" to the question "How much does this bother you?"
  A subject will be considered a surgical failure if any ONE of the criteria above is met. Otherwise, a subject will be considered a surgical success
Hospital length of stay (hours) | Up to 7 days
  Time period between hospital admission and discharge for the surgical encounter
Surgical encounter total direct costs ($) | Up to 7 days
  The costs generated by each department of the hospital involved in the surgical patient care, including hospital preoperative, intraoperative, and postoperative costs. This comprises costs related to anesthesia, surgery, operating room, medication, laboratory (including blood transfusion), equipment, and room and board.
Estimated blood loss (ml) | Day of surgery
  Mutual estimation by the surgeon and anesthesiologist
Frequency of perioperative complications (%) | 6 week
  A perioperative complication will be defined as any documented complication encountered intraoperatively through the sixth postoperative week. Complications include: visceral injury (bowel, bladder, or ureteral), need for blood transfusion, urinary tract infection (defined as patient symptoms with or without a positive urine culture that is treated with antibiotics), wound infection or abscess, readmission, and return to the operating room.
Mean Pelvic Floor Disability Index (PFDI-20) questionnaire score at the 6 week postoperative visit | 6 week
  The degree of bother and distress (quality-of-life) caused by pelvic floor symptoms is measured by the pelvic floor disability index (PFDI-20) questionnaire. The PFDI-20 has 20 items within 3 scales of symptoms (total of 20 items). Each item produces a response of 0 to 4, the average response in each scale is multiplied by 25 to obtain the scale score (range 0 to 100). The total score is the sum of the three scale score with a range of 0-300. Higher values indicate a greater degree of bother.
Mean Pelvic Floor Disability Index (PFDI-20) questionnaire score at the 6 month postoperative visit | 6 month
  The degree of bother and distress (quality-of-life) caused by pelvic floor symptoms is measured by the pelvic floor disability index (PFDI-20) questionnaire. The PFDI-20 has 20 items within 3 scales of symptoms (total of 20 items). Each item produces a response of 0 to 4, the average response in each scale is multiplied by 25 to obtain the scale score (range 0 to 100). The total score is the sum of the three scale score with a range of 0-300. Higher values indicate a greater degree of bother.
Mean Pelvic Floor Disability Index (PFDI-20) questionnaire score at the 12 month postoperative visit | 12 month
  The degree of bother and distress (quality-of-life) caused by pelvic floor symptoms is measured by the pelvic floor disability index (PFDI-20) questionnaire. The PFDI-20 has 20 items within 3 scales of symptoms (total of 20 items). Each item produces a response of 0 to 4, the average response in each scale is multiplied by 25 to obtain the scale score (range 0 to 100). The total score is the sum of the three scale score with a range of 0-300. Higher values indicate a greater degree of bother.
Mean Pelvic Floor Impact (PFIQ-7) questionnaire score at the 6 week postoperative visit | 6 week
  The life impact in women with pelvic floor disorders is measured by the pelvic floor impact (PFIQ-7) questionnaire. The PFIQ-7 consists of 7 items for each of 3 scales (total of 21 items) taken from the Urinary Impact Questionnaire, the Pelvic Organ Prolapse Impact Questionnaire, and the Colorectal-Anal Impact Questionnaire.Each item produces a response of 0 to 3, the average response in each scale is multiplied by 100/3 to obtain the scale score (range 0 to 100). The total score is the sum of the three scale score with a range of 0-300. Higher values indicate a greater degree of bother.
Mean Pelvic Floor Impact (PFIQ-7) questionnaire score at the 6 month postoperative visit | 6 month
  The life impact in women with pelvic floor disorders is measured by the pelvic floor impact (PFIQ-7) questionnaire. The PFIQ-7 consists of 7 items for each of 3 scales (total of 21 items) taken from the Urinary Impact Questionnaire, the Pelvic Organ Prolapse Impact Questionnaire, and the Colorectal-Anal Impact Questionnaire.Each item produces a response of 0 to 3, the average response in each scale is multiplied by 100/3 to obtain the scale score (range 0 to 100). The total score is the sum of the three scale score with a range of 0-300. Higher values indicate a greater degree of bother.
Mean Pelvic Floor Impact (PFIQ-7) questionnaire score at the 12 month postoperative visit | 12 month
  The life impact in women with pelvic floor disorders is measured by the pelvic floor impact (PFIQ-7) questionnaire. The PFIQ-7 consists of 7 items for each of 3 scales (total of 21 items) taken from the Urinary Impact Questionnaire, the Pelvic Organ Prolapse Impact Questionnaire, and the Colorectal-Anal Impact Questionnaire.Each item produces a response of 0 to 3, the average response in each scale is multiplied by 100/3 to obtain the scale score (range 0 to 100). The total score is the sum of the three scale score with a range of 0-300. Higher values indicate a greater degree of bother.
Mean Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) score at the 6 month postoperative visit | 6 month
  Sexual function in women with pelvic organ prolapse is measured by the PISQ-12. The scores range from 0-48 with lower scores indicating better sexual function. Scores are calculated by totalling the scores for each question with (4) always, (3) usually, (2) sometimes, (1) seldom, and (0) never. Reverse scoring is used for items 1, 2, 3 and 4. The short form questionnaire can be used with up to two missing responses. To handle missing values, the sum is calculated by multiplying the number of items by the mean of the answered items.
Mean Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) score at the 12 month postoperative visit | 12 month
  Sexual function in women with pelvic organ prolapse is measured by the PISQ-12. The scores range from 0-48 with lower scores indicating better sexual function. Scores are calculated by totalling the scores for each question with (4) always, (3) usually, (2) sometimes, (1) seldom, and (0) never. Reverse scoring is used for items 1, 2, 3 and 4. The short form questionnaire can be used with up to two missing responses. To handle missing values, the sum is calculated by multiplying the number of items by the mean of the answered items.
Mean postoperative numerical rating scale (NRS) score of pain intensity at 1 week after surgery | 1 week
  Postoperative pain is measured by the numeric rating scale (NRS 0-10; 0, no pain; 10, worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Tristi Muir, MD, Principal Investigator — The Methodist Hospital Research Institute; Danny Mounir, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No